CLINICAL TRIAL: NCT01841216
Title: EMG Activation of Gluteal Musculature and Perceived Exertion During Therapeutic Exercises With and Without Thera-Band® Resistance
Brief Title: EMG Activation of Gluteal Musculature During Exercises With and Without Resistance
Acronym: GlutEMG02
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sport and Spine Rehab Clinical Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SSR02
Record Dates: First submitted 2013-04-23; First posted 2013-04-26 (Estimated); Results first posted 2015-02-03 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-01

CONDITIONS: Low Back Pain
Keywords: Gluteus Maximus; Gluteus Medius; TFL; EMG; Perceived Exertion; Thera-Band
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Back Pain (Experimental): Lower Body Exercises with and without resistance
  Interventions: Device: Lower Body Exercises with and without resistance
- Healthy (Experimental): Lower Body Exercises with and without resistance
  Interventions: Device: Lower Body Exercises with and without resistance

INTERVENTIONS:
Device: Lower Body Exercises with and without resistance — lower body exercises with and without resistance designed to activate the gluteal/hip musculature

SUMMARY:
The gluteus medius (Gmed) and gluteus maximus (Gmax) muscles are important components in the treatment of many lower limb injuries. Recent studies have evaluated a myriad of exercises which activate the Gmed and Gmax, but limited research remains on exercises involving resistance and the role of the TFL. The purpose of this study is to evaluate Gmed, Gmax, and TFL percent maximal voluntary isometric contraction (%MVIC) and perceived exertion in healthy and low back pain patients while performing exercises with and without resistance. Methods: A convenience sample of healthy subjects and patients diagnosed with non-radicular low back pain will be recruited. Exclusionary criteria will include: current low back or lower extremity injury (healthy group), pregnancy, history of hip surgery, and radicular symptoms. Surface electromyography will be used to quantify the activity level of the gluteal muscles and TFL while performing a series of 8 exercises with and without Thera-Band® Resistance Tubing and Stability Trainer. The maximal voluntary isometric contraction (MVIC) will be established for each muscle group and the order of exercises performed will be randomized to minimize the effect of fatigue. Following the completion of each exercise, the patient will rate their perceived exertion level on the Thera-Band® Resistance Intensity Scale for Exercise (RISE). The EMG signals will be smoothed and rectified and analyzed using a root-mean-square algorithm. Clinical Relevance: The results of this study will allow clinicians to better prescribe exercises, proven to activate the gluteal muscles and limit the TFL involvement, in the treatment of low back pain.

ELIGIBILITY:
Inclusion Criteria:

* healthy, physically active subjects
* patients diagnosed with non-radicular low back pain
* 18-65

Exclusion Criteria:

* current low back or lower extremity injury (healthy group)
* pregnancy
* history of hip surgery
* radicular symptoms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barton Bishop, DPT, Principal Investigator — Sport & Spine Rehab Clinical Research Foundation
Locations (1):
- Sport & Spine Rehab, Rockville, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Back Pain | Healthy
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Back Pain | Healthy | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 15 | 14 | 29
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 36.2 [23 to 61] | 29 [18 to 47] | 32.6 [18 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 11 | 17
  Male | 9 | 4 | 13
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 11 | 11 | 22
  African American | 2 | 1 | 3
  Asian | 1 | 0 | 1
  Hispanic/Latino | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percent of Maximal Voluntary Isometric Contraction (%MVIC)
Description: Percent of Maximal Voluntary Isometric Contraction was measured by placing EMG leads on selected muscles. Data was collected and analyzed with the MyoResearch XP Masters Edition (Noraxam Inc., Scottsdale, AZ). The EMG signals were smoothed and rectified and analyzed using a root-mean-square algorithm. We used visual onset and offset of the EMG signal amplitude to select the middle 3 of 5 trials. The middle three repetitions were analyzed. Average activation and peak activation were determined and then compared to the maximum voluntary isometric contraction (MVIC), captured during a manual muscle test, for each muscle group, and expressed as a %MVIC. The %MVIC can be greater than 100% since the MVIC is captured in a stationary, isometric position using manual force and all other activities are performed in motion against elastic or gravity resistance.
Time Frame: One 40 minute session
Measure: Mean (Standard Deviation); unit: percentage of MVIC of gmax
Arm/Group | Low Back Pain | Healthy
Number analyzed (Participants) | 15 | 15
percentage of MVIC of gmax
  ClamsR | 73.5 (17.8) | 57.6 (17.8)
  Clams | 62.7 (12.6) | 37 (12.6)
  HipExt | 41.5 (8.6) | 28.6 (8.6)
  STHipExtR | 44.1 (12.3) | 23.8 (12.3)
  SLHipAB | 59.3 (12.9) | 37.2 (12.9)
  STHipAB_R | 55.8 (11.9) | 37 (11.9)
  QuadHipExt | 44.9 (8) | 23.5 (8)
  QuadHipExtR | 54.1 (12.2) | 26.5 (12.2)
  Bridge | 33.6 (7.7) | 16.9 (7.7)
  BridgeR | 37.3 (6.9) | 20.8 (6.9)
  FireHydrant | 86.4 (16) | 52.5 (16)
  FireHydrantR | 93.9 (17.3) | 57.3 (17.3)
  Lunge | 55.8 (12.8) | 25.1 (12.8)
  LungeR | 50.9 (11.9) | 24.2 (11.9)
  RunningMan | 102.5 (23.7) | 56.1 (23.7)
  RunningManR | 103.4 (21.5) | 56 (21.5)

2. Secondary Outcome: Perceived Exertion
Description: Thera-Band(R) RISE (Resistance Intensity Scale for Exercise) Scale to measure amount of perceived exertion during resistance band exercises. This is a scale 0 to 10, 0 being extremely easy and 10 being extremely hard. The subject rated the intensity or resistance felt on each exercise on this scale. The ideal range for an exercise is in the middle of the scale (4-7) where the subject is feeling resistance but is not maximally exerted.
Time Frame: 16 exercises during one 40 minute session
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Low Back Pain | Healthy
Number analyzed (Participants) | 15 | 15
units on a scale
  Clams | 1.7 [0 to 7] | 2.1 [0 to 5]
  ClamsR | 2.8 [0 to 6] | 2.9 [0 to 6]
  PrHipExt | 2.5 [0 to 8] | 2.3 [0 to 5]
  StHipExt | 3 [1 to 5] | 2.7 [0 to 6]
  SLAB | 1.5 [0 to 3] | 1.8 [0 to 4]
  StABR | 3.4 [1 to 5] | 2.2 [0 to 6]
  QHipExt | 2.3 [1 to 6] | 1.3 [0 to 3]
  QHipExtR | 3.3 [1 to 6] | 2.3 [1 to 4]
  Bridge | 1.9 [0 to 5] | 1.5 [0 to 6]
  BridgeR | 2.5 [1 to 4] | 2.1 [0 to 5]
  Fire Hydrant | 2.4 [1 to 7] | 2.3 [0 to 4]
  Fire HydrantR | 3.7 [1 to 6] | 3.2 [1 to 5]
  Lunge | 2.9 [0 to 8] | 2.2 [0 to 5]
  LungeR | 2.9 [0 to 6] | 2.7 [0 to 5]
  Running Man | 3.4 [0 to 8] | 3.2 [1 to 5]
  RunningManR | 4.4 [1 to 8] | 4.3 [1 to 6]

ADVERSE EVENTS:
Arm/Group | Low Back Pain | Healthy
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No